CLINICAL TRIAL: NCT05204888
Title: myAirvo 3 (High Flow Nasal Therapy; HFNT) for COPD Patients in the Home - a Multi-center Randomized Controlled Trial
Brief Title: myAirvo 3 (High Flow Nasal Therapy; HFNT) for COPD Patients in the Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 268447
Record Dates: First submitted 2021-12-20; First posted 2022-01-24 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients assigned to the HFNT group will be provided a myAirvo 3 device. The myAirvo 3 is a humidifier with integrated flow generator that delivers warmed and humidified respiratory gases to spontaneously breathing patients through a variety of patient interfaces. The interface used in this trial is the Optiflow™ + Duet nasal cannula sized for patient comfort. Patients will also be provided with a pulse oximetry device that connects to the myAirvo 3 to record pulse oximetry and heart rate once daily after wearing the device for two minutes.
  Patients assigned to the control group will be provided with a pulse oximetry device to record pulse oximetry and heart rate once daily after using the pulse oximeter for two minutes as well as answering a respiratory questionnaire and input data into a smartphone adapted to be used as an electronic diary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual COPD care (Active Comparator): The intervention : A pulse oximeter to record heart rate and pulse oximetry on a daily basis will be provided. A smart phone and charger will also be provided to answer a short questionnaire that queries daily respiratory symptoms plus enter heart rate and pulse oximetry data
  Interventions: Device: Pulse oximeter
- Usual COPD care with use of the myAirvo 3 integrated humidifier and flow generator. (Active Comparator): The intervention is the myAirvo 3 humidifier with integrated flow generator delivered through the Optiflow™ + Duet nasal cannula.
  Interventions: Device: myAirvo3

INTERVENTIONS:
Device: myAirvo3 — For patients assigned to the HFNT intervention group, a myAirvo 3 device will be provided. The myAirvo 3 is for the treatment of spontaneously breathing patients, infant to adult, who would benefit from receiving high flow warmed and humidified respiratory gases. This includes patients who have had upper airways bypassed. The flow may be from 2 - 60 L/min depending on the patient interface. The myAirvo 3 is for patients in homes and long-term care facilities.
  Arms: Usual COPD care with use of the myAirvo 3 integrated humidifier and flow generator.
Device: Pulse oximeter — A pulse oximeter will be provided to measure heart rate and pulse oximetry; subjects will enter and transmit the data on the smartphone once daily before 11AM. Heart rate and pulse oximetry measures will be taken after wearing the device for approximately 2 minutes.
  Arms: Usual COPD care

SUMMARY:
Parallel-group, prospective, randomized, controlled phase III trial of home High flow Nasal Therapy (HFNT) via myAirvo 3 plus usual COPD medical care vs. usual COPD medical care, for at least 1 year and up to two years in 642 GOLD Grade D, Stages II-IV patients with moderate to very severe COPD at risk for moderate and severe exacerbations with a prior history of severe exacerbation requiring hospitalization within the past 6 weeks.

DETAILED DESCRIPTION:
Objectives:

Primary Objective: To determine if HFNT delivered by myAirvo 3 increases the time to first moderate exacerbation orsevere exacerbation or all-cause mortality in patients with moderate to very severe COPD

Secondary Objectives:

To determine if HFNT delivered by myAirvo 3

1. increases the time to first severe exacerbation
2. increases the time to first exacerbation (moderate or severe)
3. reduces severe exacerbation frequency
4. reduces moderate and severe exacerbation frequency
5. reduces hospitalization duration
6. improves quality of life
7. reduces dyspnea
8. reduces PCO2
9. is safe and well tolerated
10. determine if any of the objectives are related to duration of daily HFNT use
11. Assess cost effectiveness of HFNT use

Exploratory objectives:

Develop objective definitions of exacerbations of differing levels of severity based on myAirvo 3 device or electronic diary collected measures of heart rate, respiratory rate, oxygen saturation, and dyspnea measured by modified visual analog score.

Endpoints: Primary Endpoint: The time to first moderate or severe exacerbation or all-cause mortality.

Primary Safety Endpoint: All data on adverse events, including reported to be not, possibly, probably, or definitely related to the use of myAirvo 3 device.

Secondary Endpoints:

* Rate of severe exacerbation, rate of moderate and severe exacerbations,
* Time to moderate exacerbation, time to severe exacerbation, time to moderate or severe exacerbation
* Hospitalization durations, from per visit data
* Quality of life by St George's Respiratory Questionnaire and SF-12
* Dyspnea, calculated mMRC and TDI over time
* Hours of daily HFNT use
* Impact of hours of daily HFNT use on any outcome
* PCO2
* Assess patient phenotype most likely to benefit from HFNT.
* Assess cost effectiveness of HFNT use

Exploratory endpoints:

* Development of objective definitions of exacerbations of differing levels of severity based on myAirvo 3 device or electronic diary collected measures of heart rate, respiratory rate, oxygen saturation, and dyspnea measured by modified visual analog score.
* HFNT settings (flow rate and temperature)

ELIGIBILITY:
To be eligible to participate in this study, an individual must meet all the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 30 years or greater
4. FEV1/FVC of < 70% and an FEV1 of < 80% (GOLD stages II - IV, Grade E)

   • Spirometry performed during the screening visit will be used to confirm GOLD stage. A prior spirometric test within the past 6 months can be substituted if available.
5. MRC ≥ 2 or CAT ≥ 10
6. Former smokers or current smokers and never-smokers are eligible for study inclusion

   • Current smokers must refrain from smoking when using supplemental oxygen or the myAirvo-3 device
7. History of a severe COPD exacerbation requiring hospitalization in the previous six weeks
8. COPD in a stable state after hospitalization defined as:

   * Clinically stable condition and have had no parenteral therapy for 24 hours.
   * Inhaled bronchodilators are required less than four-hourly.
   * Oxygen delivery has ceased for 24 hours (unless home oxygen is indicated).
   * If previously able, the patient is ambulating safely and independently, and performing activities of daily living.
   * The patient can eat and sleep without significant episodes of dyspnea.
   * The patient or caregiver understands and can administer medications.
   * Follow-up and home care arrangements (e.g., home oxygen, homecare, Meals on Wheels, community nurse, allied health, GP, specialist) have been completed.
9. Willing to adhere to the daily use of the myAirvo 3 regimen for at least 8 hours each day preferably at night following being shown and using the device
10. Willing to record daily symptoms and pulse oximetry and heart rate on daily basis
11. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation

    Highly effective contraception is defined as:
    * A tubal ligation:
    * An approved hormonal contraceptive such as oral contraceptives, emergency contraception used as directed, patches, implants, injections, rings or intrauterine devices
12. Able to read and communicate in English
13. Have a home environment suitable for myAirvo 3 use.
14. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration - refraining from smoking while receiving supplemental oxygen or the myAirvo-3 device

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current self-reported chronic use of positive airway pressure (PAP) therapy; continuous positive airway pressure (CPAP), or non-invasive positive pressure ventilation (NPPV)
2. A STOPBang Questionnaire score > 5*
3. Pregnancy or lactation
4. Treatment with another investigational drug or other intervention within the previous 30 days
5. Life expectancy less than 12 months due to COPD or other comorbid condition.
6. Recent upper airway surgery (within the previous month)
7. Recent head or neck trauma (within the previous month)
8. Inability to tolerate nasal prongs
9. Requirement of oxygen greater than 15 L/min

   * subjects with a STOPBang questionnaire score of > 5 may be eligible if a recent sleep study (within the previous 3 months) shows the absence of obstructive sleep apnea or the subject has, or is at risk of OSA, but refuses to use an OSA device and all other eligibility criteria are met.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To determine if myAirvo 3 use increases the time to first moderate exacerbation/severe exacerbation (hospitalization)/all-cause mortality in patients with moderate to very severe COPD. | 1 year
  Time to first moderate or severe COPD exacerbation

SECONDARY OUTCOMES:
Time to first severe exacerbation | 1 year
  To determine if HFNT delivered by myAirvo 3 increases the time to first severe exacerbation
Time to moderate or severe exacerbation | 1 year
  To determine if HFNT delivered by myAirvo 3 increases the time to first exacerbation (moderate or severe)
Severe exacerbation frequency | 1 year
  To determine if HFNT delivered by myAirvo 3 reduces severe exacerbation frequency
Moderate/severe exacerbation frequency | 1 year
  To determine if HFNT delivered by myAirvo reduces moderate and severe exacerbation frequency
Hospital length of stay | 1 year
  To determine if HFNT delivered by myAirvo 3 reduces hospitalization duration
Quality of life - SF-12 questionnaire | 1 year
  To determine if HFNT delivered by myAirvo improves quality of life as measured by the SF-12
Quality of life - Severe Respiratory Insufficiency Questionnaire | 1 year
  To determine if HFNT delivered by myAirvo improves quality of life as measured by the Severe Respiratory Insufficiency Questionnaire
Quality of life - Saint George's Respiratory Questionnaire | 1 year
  To determine if HFNT delivered by myAirvo improves quality of life as measured by the Saint George's Respiratory Questionnaire
Quality of life - Baseline Dyspnea Index and Transitional Dyspnea Index | 1 year
  To determine if HFNT delivered by myAirvo improves quality of life as measured by the EQ-5D questionnaire
Dyspnea | 1 year
  To determine if HFNT delivered by myAirvo reduces dyspnea as measured by the Baseline Dyspnea Index and Transitional Dyspnea Index
pCO2 reduction | 1 year
  To determine if HFNT delivered by myAirvo reduces pCO2
Adverse event reporting | 1 year
  To determine if HFNT delivered by myAirvo is safe and well tolerated
Correlations with average hours of use | 1 year
  To determine if any of the above outcomes are related to duration of daily HFNT use
Cost effectiveness | 1 year
  To assess the cost effectiveness of HFNT use in COPD

CONTACTS AND LOCATIONS:
Locations (27):
- United States (25):
  - UAB School of Medicine/Lung Health Center, Birmingham, Alabama
  - Honor Health, Scottsdale, Arizona
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Alloy Clinical Research, Kissimmee, Florida
  - Reliable Research, Inc., Miami, Florida
  - NewGen Health Group, Miami, Florida
  - Destiny Research, Palmetto Bay, Florida
  - University of Chicago, Chicago, Illinois
  - The Iowa Clinic, West Des Moines, Iowa
  - University of Maryland - Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Clinical Research Associates of Central Pennsylvania, DuBois, Pennsylvania
  - Jeanes Hospital, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - The University of Pittsburgh, Pittsburgh, Pennsylvania
  - Respire Research Institute, Houston, Texas
  - The University of Vermont Medical Center, Inc, Burlington, Vermont
  - West Virginia Clinical and Translational Science Institute, Morgantown, West Virginia
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - The Research Institute of McGill University Health Centre, Montreal, Quebec City

IPD SHARING:
Plan to Share IPD: No